CLINICAL TRIAL: NCT05969886
Title: Predictive Value of Ventricular-Arterial Coupling for Post-Induction Hypotension: A Prospective Observational Cohort Study
Brief Title: Ventricular-Arterial Coupling: A Predictor of Post-Induction Hypotension
Acronym: VAC
Status: Completed | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 32/GCN-HDDD; No: 32/GCN-HDDD (Other: University Medical Center Ho Chi Minh City)
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Hypotension on Induction
Keywords: Ventricular-Arterial Coupling (VAC); Ea/Ees ratio; Post-induction hypotension (PIH); Risk factors for PIH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-induction hypotension (PIH) is a common occurrence during the period from induction of general anesthesia to initiation of incision. PIH has been identified as an independent risk factor for postoperative major complications. Identifying high-risk patients for PIH could potentially help prevent its occurrence. Several risk factors associated with PIH have been identified, including patient conditions and use of specific anesthetic agents. Ventricular-arterial coupling (VAC) is evaluated using the ratio Ea/Ees and represents the interaction between the left ventricle (LV) and the arterial system. It reflects how changes in LV contractility (Ees) and changes in arterial load (Ea) work together to maintain optimal LV performance. A study aims to investigate the relationship between preoperative Ea/Ees ratio and the incidence of PIH (defined as MAP < 65 mmHg).

DETAILED DESCRIPTION:
Post-induction hypotension (PIH) is a common event due to general anesthesia in patients undergoing surgery. It is described as hypotension occurring during the period from induction of general anesthesia to initiation of incision. A universal definition of intraoperative hypotension is lacking, leading to inconsistent rates of occurrence for PIH. According to Yoshimura et al., PIH occurs in 34% of patients using the mean arterial pressure (MAP) definition of < 55 mmHg, whereas Maheshwari found PIH in 53% of patients using a MAP definition of < 65 mmHg. Furthermore, Maheshwari et al. demonstrated that PIH was an independent risk factor for postoperative major complications such as myocardial injury, cerebrovascular events, and acute kidney injury.

If high-risk patients for PIH could be identified we might potentially prevent PIH. In a systematic review, Chen et al. pointed out that the risk factors associated with PIH were ASA (American Society of Anesthesiologists) III-V, advanced age, emergency cases, hypovolaemia, long-term use of angiotensin-converting enzyme inhibitors or angiotensin receptor blockers, use of propofol and high-dose of opioid. This study suggests that PIH may be the result of an interaction between the anesthetic agent and the cardiovascular condition of the patient. Conditions such as moderate-to-severe aortic regurgitation, moderate-to-severe mitral regurgitation, regional wall motion abnormalities, and echocardiography findings (e.g. elevated ratio of peak early diastolic transmitral flow velocity to annular velocity) have been identified as PIH-independent risk factors.

End-systolic elastance (Ees) is a measure of the contractile state of the left ventricle (LV). It represents the relationship between LV end-systolic pressure (LVESP) and end-systolic volume (ESV). Effective arterial elastance (Ea) is a measure of the total arterial load on the LV and is calculated as the ratio of LVESP to stroke volume (SV). Ventricular-arterial coupling (VAC), assessed by the ratio Ea/Ees, describes the interaction between the LV and arterial system. VAC reflects the interplay between the changes in LV contractility (Ees) and changes in arterial load (Ea) to maintain optimal LV performance.

Aktas et al. analyzed Ea as a predictor of PIH. The results of this study showed that pre-induction Ea had excellent predictability of hypotension. However, Ees values were not determined, thus making it speculative to conclude that pre-induction VAC is impaired in patients with high Ea. There are no studies available that assessed the role of preoperative VAC in predicting PIH. Therefore, we will investigate the relationship between the preoperative Ea/Ees ratio and the incidence of PIH (: hypotension being defined as MAP < 65 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* Patients with ASA (American Society of Anesthesiologists) physical status 1 - 4.
* Elective surgery.
* Preoperative transthoracic echocardiography was performed within 48 hours before surgery. The values of Ees and Ea were determined by the method of Chen.
* Patients consented to participate in the study.
* Patients scheduled for surgery undergoing standard general anesthesia (protocol: see below) with endotracheal intubation.
* Patients were hemodynamically stable until the preoperative period.

Exclusion Criteria:

* Cardiac and obstetric surgery.
* Allergy to any anesthetic drug.
* Arrhythmia.
* Severe valvular heart disease.
* Severe pre-existing lung disease.
* Mean pulmonary arterial pressure (PAPm ≥ 40 mmHg).
* Anticipation of difficult airway management.
* Hypotension occurs during the induction of anesthesia due to suspected anaphylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with American Society of Anesthesiologists (ASA) physical status 1 - 4 who underwent elective surgery
Sampling Method: Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Prediction | from induction of anesthesia to incision initiation
  Investigate the predictive value of the Ea/Ees ratio (along with echocardiographic variables) on PIH.

SECONDARY OUTCOMES:
Incidence | from induction of anesthesia to incision initiation
  Determine the frequency of PIH

CONTACTS AND LOCATIONS:
Overall Officials: Khoi M Le, Assoc.Prof, Study Director — University Medical Center
Locations (1):
- University Medical Centre Ho Chi Minh, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Yes, there is a plan to make individual participant data (IPD) available. The de-identified dataset underlying the findings of this study will be shared upon reasonable request. Researchers can request access by contacting chinh.lh@umc.edu.vn. Requests will be reviewed to ensure compliance with ethical and legal standards.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the study. Indefinitely
Access Criteria: "Data will be shared upon reasonable request, with approval based on the researcher's qualifications and the purpose of the request." Access will only be granted to academic or non-commercial researchers who meet the conditions outlined in the Data Use Agreement.

REFERENCES:
- [Result] Yoshimura M, Shiramoto H, Koga M, Morimoto Y. Preoperative echocardiography predictive analytics for postinduction hypotension prediction. PLoS One. 2022 Nov 28;17(11):e0278140. doi: 10.1371/journal.pone.0278140. eCollection 2022. PMID 36441797
- [Result] Maheshwari K, Turan A, Mao G, Yang D, Niazi AK, Agarwal D, Sessler DI, Kurz A. The association of hypotension during non-cardiac surgery, before and after skin incision, with postoperative acute kidney injury: a retrospective cohort analysis. Anaesthesia. 2018 Oct;73(10):1223-1228. doi: 10.1111/anae.14416. Epub 2018 Aug 24. PMID 30144029
- [Result] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066
- [Result] Chen B, Pang QY, An R, Liu HL. A systematic review of risk factors for postinduction hypotension in surgical patients undergoing general anesthesia. Eur Rev Med Pharmacol Sci. 2021 Nov;25(22):7044-7050. doi: 10.26355/eurrev_202111_27255. PMID 34859868
- [Result] Tarao K, Daimon M, Son K, Nakanishi K, Nakao T, Suwazono Y, Isono S. Risk factors including preoperative echocardiographic parameters for post-induction hypotension in general anesthesia. J Cardiol. 2021 Sep;78(3):230-236. doi: 10.1016/j.jjcc.2021.03.010. Epub 2021 Apr 8. PMID 33838982
- [Result] Monge Garcia MI, Santos A. Understanding ventriculo-arterial coupling. Ann Transl Med. 2020 Jun;8(12):795. doi: 10.21037/atm.2020.04.10. PMID 32647720
- [Result] Guinot PG, Andrei S, Longrois D. Ventriculo-arterial coupling: from physiological concept to clinical application in peri-operative care and ICUs. Eur J Anaesthesiol Intensive Care. 2022 Aug 3;1(2):e004. doi: 10.1097/EA9.0000000000000004. eCollection 2022 Apr. PMID 39916686
- [Result] Aktas Yildirim S, Sarikaya ZT, Dogan L, Ulugol H, Gucyetmez B, Toraman F. Arterial Elastance: A Predictor of Hypotension Due to Anesthesia Induction. J Clin Med. 2023 Apr 27;12(9):3155. doi: 10.3390/jcm12093155. PMID 37176595
- [Result] Chen CH, Fetics B, Nevo E, Rochitte CE, Chiou KR, Ding PA, Kawaguchi M, Kass DA. Noninvasive single-beat determination of left ventricular end-systolic elastance in humans. J Am Coll Cardiol. 2001 Dec;38(7):2028-34. doi: 10.1016/s0735-1097(01)01651-5. PMID 11738311
- [Result] Mitchell C, Rahko PS, Blauwet LA, Canaday B, Finstuen JA, Foster MC, Horton K, Ogunyankin KO, Palma RA, Velazquez EJ. Guidelines for Performing a Comprehensive Transthoracic Echocardiographic Examination in Adults: Recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2019 Jan;32(1):1-64. doi: 10.1016/j.echo.2018.06.004. Epub 2018 Oct 1. No abstract available. PMID 30282592
- [Result] Cho JY, Kim KH. Evaluation of Arterial Stiffness by Echocardiography: Methodological Aspects. Chonnam Med J. 2016 May;52(2):101-6. doi: 10.4068/cmj.2016.52.2.101. Epub 2016 May 20. PMID 27231673
- [Result] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963
- [Result] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600